CLINICAL TRIAL: NCT01894724
Title: Targeted Cerebral Hypothermia During Cardiac Surgery: A Feasibility Trial
Brief Title: Targeted Hypothermia During Cardiac Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroSave Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-1.0
Record Dates: First submitted 2013-06-30; First posted 2013-07-10 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NeuroSave Device (Experimental): Targeted Hypothermia with NeuroSave Device
  Interventions: Device: NeuroSave device

INTERVENTIONS:
Device: NeuroSave device

SUMMARY:
This study designed to evaluate the safety and feasibility of the NeuroSave device to rapidly reduce brain temperature while maintaining the brain at a lower temperature than the body core during cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Undergoing coronary revascularization or valvular cardiac surgery
* The study patient or the study patient's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Human Research Ethics Committee (HREC) of the respective clinical site
* The study patient agrees to comply with all study -related procedures

Exclusion Criteria:

* Women known or suspected to be pregnant (as confirmed by a pregnancy test for all women of child-bearing age)
* Past history of cerebrovascular accident (stroke or TIA)
* History of clinically diagnosed active psychiatric conditions
* Emergency or salvage cardiac valve operations
* Body weight < 50 kg
* Leukopaenia (WBC < 3000 cell/mL), anaemia (Hgb < 11g/dL), Thrombocytopaenia (Plt < 50,000 cell/mL)
* Active upper GI bleeding within 3 months (90 days) prior to procedure
* Renal insufficiency (creatinine > 265 micromol/L) and/or renal replacement therapy at the time of screening
* Estimated life expectancy < 12 months (365 days)
* Structural abnormality or disease of nose, mouth, pharynx and oesophagus (excluding gastric reflux oesophagus disease),
* Currently participating in an investigational drug or another device study that would potentially impact the results of this study as determined by the PI. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Freedom from major adverse events related to the use of the NeuroSave device | Surgery through discharge (up to 5 days post-surgery)

SECONDARY OUTCOMES:
Brain-core temperature differential during cardiac surgery | Continuously assessed over course of cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Silvanna Marasco, Principal Investigator — The Alfred
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia